CLINICAL TRIAL: NCT05056870
Title: Clinical Evaluation of Spherical Soft Contact Lenses, Toric Soft Contact Lenses and Spectacles in Low Astigmats
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6459
Record Dates: First submitted 2021-09-15; First posted 2021-09-27 (Actual); Results first posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test/Control (Experimental): Eligible subjects will be randomized to the sequence, Test/Control
  Interventions: Device: ACUVUE Oasys 1-Day with HydraLuxe Technology for Astigmatism; Device: ACUVUE Oasys 1-Day with HydraLuxe Technology
- Control/Test (Experimental): Eligible subjects will be randomized to the sequence, Control/Test
  Interventions: Device: ACUVUE Oasys 1-Day with HydraLuxe Technology for Astigmatism; Device: ACUVUE Oasys 1-Day with HydraLuxe Technology

INTERVENTIONS:
Device: ACUVUE Oasys 1-Day with HydraLuxe Technology for Astigmatism — TEST
Device: ACUVUE Oasys 1-Day with HydraLuxe Technology — CONTROL

SUMMARY:
This will be a 5-visit, randomized, partially single-masked, bilateral wear, dispensing, 2-treatment × 2-period crossover study with spectacle-wear washout and wash-in periods.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy of all the following criteria to be enrolled in the study.

  1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Be between 18 and 39 (inclusive) years of age at the time of screening.
  4. By self-report, habitually wear soft contact lenses (sphere or toric) in both eyes in a daily reusable or daily disposable wear modality (i.e. not extended wear modality). Habitual wear is defined as a minimum of 6 hours of wear per day, for a minimum of 2 days per week during the past 4 weeks.
  5. Possess a wearable pair of spectacles that provide correction for distance vision.
  6. In both eyes, have magnitude of the cylinder component of their vertex-corrected distance refraction greater than or equal to 0.625 DC and less than 1.625 DC.
  7. In both eyes, have the mean sphere of their vertex-corrected distance refraction minus half of the indicated contact lens label cylinder power be between -0.875 to -4.625 DS (inclusive).
  8. For each eye, have the cylinder axis of their distance refraction between 165° and 15° (i.e., 180±15°, inclusive) or between 75° and 105° (i.e., 90±15°, inclusive).
  9. For both eyes, have the sphere power of their habitual spectacles within ±0.50 Diopters Sphere (DS) (inclusive) of the sphere power of their current subjective refraction.
  10. For both eyes, have the cylinder power of their habitual spectacles within ±0.50 Diopters Cylinder (DC) (inclusive) of the cylinder power of their current subjective refraction.
  11. For both eyes, have the cylinder axis of their habitual spectacles within ±20° (inclusive) of the cylinder axis of their current subjective refraction.
  12. Achieve monocular VA of 20/30 or better with their habitual spectacles in both eyes.

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Be currently pregnant or lactating.
  2. Be diabetic.
  3. Be currently using any ocular medications or have any ocular infection of any type.
  4. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g. rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See section 9.1 for additional details regarding excluded systemic medications.
  5. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 6 months.
  6. Be currently wearing monovision or multifocal contact lenses.
  7. Be currently wearing lenses in an extended wear modality.
  8. Have a history of strabismus or amblyopia.
  9. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
  10. Have participated in a contact lens or lens care product clinical trial within 7 days prior to study enrollment.
  11. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
  12. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
  13. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (13):
- United States (13):
  - Eyecenter Optometric, Rocklin, California
  - Sabal Eye Care, Longwood, Florida
  - Maitland Vision Center, Maitland, Florida
  - Windward Vision Ctr Associates Inc., Kaneohe, Hawaii
  - Indiana University School of Optometry, Bloomington, Indiana
  - Advanced Eye Care, Raytown, Missouri
  - Sacco Eye Group, Vestal, New York
  - University Hospitals of Cleveland Medical Center, Cleveland, Ohio
  - ProCare Vision Center, Granville, Ohio
  - Professional Visioncare Inc., Westerville, Ohio
  - Total Eye Care, Memphis, Tennessee
  - Tyler Texas Associates, Tyler, Texas
  - Botetourt Eyecare, LLC, Salem, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 174 subjects were enrolled in this study. Of those enrolled, a total of 161 subjects were assigned to one of two wear sequences; while 13 subjects were screen failure and/or not assigned. Of the total assigned subjects, 151 subjects completed the study while, 10 subjects were discontinued from the study.
Groups:
- Test/Control: Subjects that wore the Test lens during Period 1 and the Control lens during Period 2.
- Control/Test: Subjects that wore the Control lens during Period 1 and the Test lens during Period 2.
Period: Period 1
Arm/Group | Test/Control | Control/Test
Started | 80 | 81
Completed | 76 | 77
Not Completed | 4 | 4
Not completed — Site COVID-19 Related | 3 | 3
Not completed — Subject Withdrawn by PI due to Non Compliance to Protocol | 0 | 1
Not completed — Subject No Longer Meets Eligibility Criteria | 1 | 0
Period: Period 2
Arm/Group | Test/Control | Control/Test
Started | 76 | 77
Completed | 74 | 77
Not Completed | 2 | 0
Not completed — COVID-19 Related | 1 | 0
Not completed — Subject No Longer Meets Eligibility Criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Subjects that wore either Test lens or Control during the study.
Arm/Group | Total
Number analyzed (Participants) | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.9 (5.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109
  Male | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 4
  Black or African American | 11
  White | 122
  More than one race | 9
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 161

OUTCOME MEASURES:

1. Primary Outcome: High Luminance High Contrast Monocular Visual Acuity (LogMAR)
Description: Visual Acuity was collected for each subject eye at distance (4 meter) using a Logarithm of Minimal Angle of Resolution (logMAR) visual acuity scale. This was evaluated under high luminance and high contrast conditions (HLHC) at 4 meters from Early Treatment Diabetic Retinopathy Study (ETDRS) charts at the 1-week follow-up visit. A value of 0.0 logMAR is equivalent to 20/20 Snellen Visual Acuity. Lower values of visual acuity indicate better vision. The average logMAR Visual Acuity was reported for each lens type.
Time Frame: 1-Week Follow-up
Population: All randomized subjects regardless of actual treatment and subsequent withdrawal from the study or deviation from the protocol. At least one observation was recorded.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Groups:
- Test (AO1DfA): Subjects that wore the Test lens during the study.
- Control (AO1D): Subjects that wore the Control lens during the study.
Arm/Group | Test (AO1DfA) | Control (AO1D)
Number analyzed (Participants) | 154 | 152
Number analyzed (eyes) | 308 | 304
logMAR | -0.126 (0.0798) | -0.028 (0.1123)
Statistical Analysis 1: Comparison: Test (AO1DfA) vs Control (AO1D); Test type: Superiority — Superiority was declared if the upper limit of the 95% confidence interval of was below 0.00 logMAR; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Mean Difference = -0.097, 95% CI 2-sided [-0.113 to -0.081], Standard Error of Mean 0.0080 — Mean difference was calculated as Test - Control

2. Secondary Outcome: CLUE Vision Score
Description: CLUE Vision Score was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average CLUE vision score for each lens type was reported.
Time Frame: 1-Week Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test (AO1DfA) | Control (AO1D)
Number analyzed (Participants) | 154 | 152
units on a scale | 69.39 (20.151) | 41.49 (28.139)
Statistical Analysis 1: Comparison: Test (AO1DfA) vs Control (AO1D); Test type: Superiority — Superiority was declared if the lower limit of the 95% confidence interval of was above 0; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Mean Difference = 28, 95% CI 2-sided [22.6 to 33.3], Standard Error of Mean 2.69 — Mean difference was calculated as Test - Control

3. Secondary Outcome: High Luminance High Contrast Monocular Visual Acuity (LogMAR)
Description: Visual Acuity was collected for each subject eye at distance (4 meter) using a Logarithm of Minimal Angle of Resolution (logMAR) visual acuity scale. This was evaluated under high luminance and high contrast conditions (HLHC) at 4 meters from Early Treatment Diabetic Retinopathy Study (ETDRS) charts at the 1-week follow-up visit. A value of 0.0 logMAR is equivalent to 20/20 Snellen Visual Acuity. Lower values of visual acuity indicate better vision. The average logMAR Visual Acuity was reported for each lens type. Data summaries for the Control lens are reported for the first primary measure outcome.
Time Frame: 1-Week Follow-up
Population: All subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Groups:
- Spectacles: Subjects that wore their own Spectacles during the wash-in period at 1-week follow-up.
Arm/Group | Test (AO1DfA) | Spectacles
Number analyzed (Participants) | 151 | 151
Number analyzed (eyes) | 302 | 302
logMAR | -0.128 (0.0799) | -0.107 (0.0812)
Statistical Analysis 1: Comparison: Test (AO1DfA) vs Spectacles; Test type: Non-Inferiority — Non-Inferiority was declared if the upper limit of the 95% confidence interval of was below 0.05 logMAR; Linear Mixed Model; Kenward and Roger method was used for denominator degrees of freedom; Mean Difference = -0.020, 95% CI 2-sided [-0.032 to -0.008], Standard Error of Mean 0.0061 — Mean difference was calculated as Test - Control

4. Secondary Outcome: Subjective Contact Lens Preference
Time Frame: 1-Week Follow-up
Population: as for outcome 1
Measure: Number; unit: proportion of participants
Arm/Group | Total
Number analyzed (Participants) | 151
proportion of participants
  Prefer Test | 0.689
  Prefer Control | 0.225
  No Preference | 0.086
Statistical Analysis 1: Comparison: Total; Test type: Superiority — Superiority was declared if the lower limit of the 95% confidence interval of was above 1; Generalized Linear Mixed Model; Mean Ratio = 2.98, 95% CI 2-sided [1.73 to 5.11] — Mean Ratio was calculated as Test over Control

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; The study duration for each subject was approximately 2 weeks.
Groups:
- Test: Subjects that wore the Test lens during either period of the study
- Control: Subjects that wore the Control lens during either period of the study.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/157 | 0/157
Serious Adverse Events (participants affected / at risk) | 0/157 | 0/157
Other Adverse Events (participants affected / at risk) | 0/157 | 0/157

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/70/NCT05056870/Prot_SAP_000.pdf